CLINICAL TRIAL: NCT02303964
Title: Pre-Hospital Use of Plasma for Traumatic Hemorrhage
Acronym: PUPTH
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low patient enrollment is the primary reason
Sponsor: Virginia Commonwealth University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM14813; IND #15910 (Registry Identifier: FDA); W81XWH-12-2-0022 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-10-06; First posted 2014-12-01 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Shock, Hemorrhagic
Keywords: Trauma; Hemorrhage; Plasma; Shock; Polytrauma
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries; Hemorrhage; Shock; Multiple Trauma | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Type A Thawed Plasma (Active Comparator): Eligible subjects with polytrauma (PT) and major hemorrhage (MH) will be randomized to receive 2 units of thawed Type A plasma in the pre-hospital setting administered by EMS first responders.
  An exception from informed consent under 21CFR 50.24 is required since enrollment will occur (for the majority of subjects) before consent can be obtained.
  Interventions: Biological: Plasma
- Normal saline (Placebo Comparator): Eligible subjects with polytrauma (PT) and major hemorrhage (MH) will be randomized to receive normal saline in the pre-hospital setting administered by EMS first responders. Normal saline is standard of care
  Interventions: Drug: Normal saline

INTERVENTIONS:
Biological: Plasma — Type A thawed plasma (up to 2 units) will be administered to polytrauma subjects randomized to plasma arm of study
  Other Names: Thawed Plasma
  Arms: Type A Thawed Plasma
Drug: Normal saline — Normal saline will be administered to polytrauma subjects randomized to normal saline arm of study
  Other Names: 0.9% Normal Saline
  Arms: Normal saline

SUMMARY:
Type A Thawed Plasma (TP) will be compared in polytrauma patients who receive only Normal Saline (NS) (standard of care) before arrival at the hospital.

The purpose of this study is to determine if prehospital administration of thawed plasma can reduce mortality of patients who have lost a large amount of blood due to their injuries, compared to those receiving standard of care.

DETAILED DESCRIPTION:
INVESTIGATIONAL PLAN This will be an open-label, non-blinded, randomized clinical trial to investigate mortality (30 days) and morbidity of Type A thawed Plasma (TP) versus NS infusion at earliest contact, administered by Emergency Medical Service (EMS) supervisors to subjects who have sustained severe Polytrauma / Major hemorrhage (PTr / MH). The total study is expected to last 2 years with 210 patients enrolled.

The two EMS agencies involved in the study will each have one EMS supervisor quick-response vehicle (QRV) equipped with an approved, validated refrigeration unit for TP transport. EMS personnel trained in plasma administration and recognition of reactions may administer up to 2 units of TP to subjects approved for study enrollment. Blood samples for coagulation and lipid testing will be drawn prior to TP administration by EMS personnel,and repeated by hospital personnel at 30 minutes, 8 hours, and 24 hours post-injury.

This study is approved for "Exception from Informed Consent" (EFIC). Once the patient has reached VCUMC and has been entered into the VCUMC health care system, the treating team will advise the Study Coordinator (SC) whether or not a subject is able to consent. As the plasma administration will occur in the field prior to arrival to VCUMC, the SC will make every effort possible to obtain consent from the subject or legally authorized representative (LAR) for continued study participation before the next intervention (8 hour blood specimen collection). The attempts to contact the LAR will be documented in detail. If a subject lacks the ability to provide his/her own consent by the end of day 30, the consent signed by the LAR will be the consent document in force at the subject's completion of the study and no further consent will be sought.

ELIGIBILITY:
Inclusion Criteria:

* Blunt or penetrating trauma,
* Blood Pressure (BP) systolic <70 mmHg or BP 70-90 mmHg with Heart Rate (HR) > 108 Beats Per Minute (BPM),
* Ongoing hemorrhage with unstable vital signs

Exclusion Criteria:

* Wearing opt-out wrist band,
* Wearing medical alert jewelry / bracelet, etc. indicating Jehovah Witness or similar with objections to blood transfusions,
* Refusal to participate (by subject or LAR),
* Communication barrier at the time of eliciting refusal (non-English speaking or non-Spanish speaking),
* Not expected to survive transport to Virginia Commonwealth University Medical Center (VCUMC),
* Documented Do Not Resuscitate (DNR) order found,
* Cardiac arrest or Cardio-Pulmonary Resuscitation (CPR) prior to randomization
* Penetrating head trauma,
* Known / obvious pregnancy,
* Prisoner,
* Burns > 20% of body surface

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 day
  all cause mortality

SECONDARY OUTCOMES:
Coagulation function (thromboelastography, RoTEM, Hemodyne, fibrinogen, D-dimer, PFA-100, platelet count, flow cytometry) | 24 hours
  thromboelastography, RoTEM, Hemodyne, fibrinogen, D-dimer, PFA-100, platelet count, flow cytometry
Vital signs (blood pressure, pulse, temperature) | 24 hours
  blood pressure, pulse, temperature
Blood product utilization (number of red blood cell units, number of plasma units, number of platelet units cryoprecipitate doses) | 30 days
  number of red blood cell units, number of plasma units, number of platelet units cryoprecipitate doses
Lipidomic profiles (arachidonic acid, eicosinoid expression, prostacyclin expression) | 24 hours
  arachidonic acid, eicosinoid expression, prostacyclin expression
Blood biochemistry (pH, bicarbonate, lactate) | 24 hours
  pH, bicarbonate, lactate
Hematology (Hemoglobin, hematocrit) | 24 hours
  Hemoglobin, hematocrit
Hospital outcomes (number of cases of multi-system organ failure (MSOF), renal failure, length of hospital stay, length of ICU stay, number of days on a ventilator, number of surgeries, number of infections) | 30 days
  number of cases of multi-system organ failure (MSOF), renal failure, length of hospital stay, length of ICU stay, number of days on a ventilator, number of surgeries, number of infections

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Spiess, MD, FAHA, Principal Investigator — VCU
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no data to share.

REFERENCES:
- [Derived] Reynolds PS, Michael MJ, Spiess BD. Application of Incident Command Structure to clinical trial management in the academic setting: principles and lessons learned. Trials. 2017 Feb 9;18(1):62. doi: 10.1186/s13063-016-1755-9. PMID 28183347
- [Derived] Reynolds PS, Michael MJ, Cochran ED, Wegelin JA, Spiess BD. Prehospital use of plasma in traumatic hemorrhage (The PUPTH Trial): study protocol for a randomised controlled trial. Trials. 2015 Jul 30;16:321. doi: 10.1186/s13063-015-0844-5. PMID 26220293